CLINICAL TRIAL: NCT04294589
Title: Evaluation of Neutrophil Extracellular Traps (NETs) by Flow Cytometry in Patients With Solid Cancers Associated With a High Risk of Venous Thromboembolic Events
Brief Title: Evaluation of NETs in Patients With Solid Cancers Associated With a High Risk of Venous Thromboembolic Events
Acronym: Flownet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190640
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer; Gastric Cancer; Colorectal Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous Thromboembolic Events (ETVs) are the second leading cause of death (9.2% of causes of death) in cancer patients after tumor progression (1). Indeed, cancer is associated with a 4 to 7-fold risk of ETV during chemotherapy (2). This complication is observed in 20% of cancer patients (3), and is sometimes an inaugural manifestation of cancer. This risk is particularly increased during the first 3 months after cancer diagnosis (4).

A biomarker correlated with the occurrence of ETVs would make it possible to target patients at high risk of thrombosis who could benefit from primary thromboprophylaxis, thus avoiding the complications, particularly haemorrhagic, and the additional costs associated with the long-term diagnostic and therapeutic management of ETVs. The investigator has implemented in the laboratory an innovative approach to the detection and quantification of circulating NETs by flow cytometry (FCM) allowing the routine determination of NETs. Therefore the investigator propose to assess NETs by CMF in a cohort of cancer patients with a very high risk of ETVs (pancreatic cancer, gastric cancer and colon cancer).

DETAILED DESCRIPTION:
The NETs will be detected and quantified by CMF on the remaining EDTA tube collected to perform the blood count (NFS), using the method in place in the laboratory, adapted from the method initially described by Gavillet et al. The analyses will be carried out on a Fortessa LSR cytometer (Becton Dickinson), the antibodies used are specific to NET components: citrullinated H3 anti-histone in indirect labelling coupled APC, PE myeloperoxidase and Hoescht 34580 as DNA marker. The level will be measured in NETs/µL of whole blood as a function of the white blood cell count (Sysmex XN-3000). In parallel, other parameters associated with ETV risk will be evaluated: NFS on Sysmex-XN PLC, D-dimers, FVIII and MP. The assays of PM, D-dimers and FVIII will be performed specifically as part of the project, the other parameters will be measured as part of routine patient management and will not result in any additional constraints or costs. Biomarker assays will be performed at the time of cancer diagnosis on the EDTA and citrate tubes collected for NFS and TP/TCA respectively as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18 years of age (≥18),
* Patient with pancreatic, gastric or colorectal cancer,
* Patient with a high risk of ETV,
* Patient on the first line of treatment or relapsing after a period of complete remission,
* Patient affiliated to a social security system or CMU.

Exclusion Criteria:

* Patient who has had an ETV in the 3 months prior to inclusion,
* Patient with a life expectancy of less than 3 months,
* Patient with an anticoagulation placement,
* Known pregnant or breastfeeding woman,
* Patient under guardianship or curatorship.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with pancreatic, gastric or colorectal cancer at high risk of ETV, on the first line of treatment or relapsing after a period of complete remission.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Show that the NETs rate is higher at diagnosis in solid cancer patients with ETV within 4 months of diagnosis compared to patients without ETV | 16 months
  At the end of the study, after a minimum clinical follow-up of 4 months, the frequency of ETVs will be correlated to the NET rate measured in univariate and multivariate analysis (including also the following thrombotic risk factors: neutrophil levels, platelet levels, D-dimers, factor VIII, procoagulant activity of PM and body mass index).

SECONDARY OUTCOMES:
Determine a threshold of NETs that optimizes management based on the consequences of classification errors through decision analysis | 16 months
  The choice of an optimal threshold of NETs (sensitivity, specificity, likelihood ratio) will be determined by decision analysis using a decision tree combining probabilities of events and costs associated with fair (true positive, true negative) and erroneous (false positive, false negative) decisions.
Explore the possibility of a prognostic VTE score integrating the NET rate and other clinical and biological parameters measured at the time of cancer diagnosis | 16 months
  The choice of an optimal threshold of NETs (sensitivity, specificity, likelihood ratio) will be determined by decision analysis using a decision tree combining probabilities of events and costs associated with fair (true positive, true negative) and erroneous (false positive, false negative) decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BARDET, PhD, Principal Investigator — hematology immunology transfusion Service, Ambroise Pare hospital
Locations (1):
- Ambroise Pare Hospital, Boulogne-Billancourt, Haut de Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khorana AA, Francis CW, Culakova E, Kuderer NM, Lyman GH. Thromboembolism is a leading cause of death in cancer patients receiving outpatient chemotherapy. J Thromb Haemost. 2007 Mar;5(3):632-4. doi: 10.1111/j.1538-7836.2007.02374.x. No abstract available. PMID 17319909
- [Background] Chew HK, Wun T, Harvey D, Zhou H, White RH. Incidence of venous thromboembolism and its effect on survival among patients with common cancers. Arch Intern Med. 2006 Feb 27;166(4):458-64. doi: 10.1001/archinte.166.4.458. PMID 16505267